CLINICAL TRIAL: NCT05356624
Title: Effects of Mobilization With Movement Versus Soft Tissue Mobilization on Pain Function and ROM in Patients With De Quervain Tenosynovitis: A Randomised Controlled Trail
Brief Title: Mobilization With Movement Versus Soft Tissue Mobilization in Patients With De Quervain Tenosynovitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0108 Ayesha
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: De Quervain Syndrome
Keywords: de quervains tenosynovitis; pain; manual therapy; ROM
MeSH Terms: conditions — De Quervain Disease; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization (Experimental): Mobilization with movement (3 sets per 10 repetitions).
  Interventions: Other: Mulligan Mobilization
- Soft tissue mobilization (Experimental): Soft tissue mobilization (3 sets per 10 repetitions)
  Interventions: Other: Soft Tissue Mobilization

INTERVENTIONS:
Other: Mulligan Mobilization — It is technique in which passive mobilization is applied by therapist to improve the normal position and by holding the passive glide active movement in restricted direction of motion to reduce pain or improve range of motion or function. A total of 3 sets of 10 repetition three times a week on alternate days for 6 week
  Arms: Mulligan Mobilization
Other: Soft Tissue Mobilization — in this technique for joint the passive glides are applied, for CMC joint mobilization patient hand is rest on table. The therapist grasp trapezium with one hand and 1st metacarpal between index and thumb of other hand to apply glide. A total of 3 sets of 10 repetition three times a week on alternate days for 6 weeks.
  Arms: Soft tissue mobilization

SUMMARY:
this study will investigate the effects of mobilization with movement in addition to soft tissue mobilization on pain and range of motion in patients suffering from De Quervain Tenosynovitis.

DETAILED DESCRIPTION:
De quervain tenosynovitis also known as stenosing tenosynovitis is a condition which occur when tendons at the base of thumb pinched and become irritated. Several treatment options are available like ultrasound, Graston therapy, thrust or non-thrust manipulation, mobilization with movement, soft tissue mobilization but this study focus on 2 treatments to improve malalignment of the joint and also reduce pain. First treatment is mobilization with movement in which passive accessory mobilization from therapist while active mobility is performed by patient. Second technique is soft tissue mobilization in which passive glides are applied. The purpose of study is to make comparison between mobilization with movement and soft tissue mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female

  * 20 to 50 years
  * Subjects with pain in base of thumb (9)
  * Subject with positive fienklstein test

Exclusion Criteria:

* History of radiculopathy

  * History of systemic illness
  * History of connective tissue disorder
  * Rheumatoid arthritis
  * History of hand or wrist injury or acute trauma
  * Subject with negative fienklstein test

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 3 months
  It is a 100 mm scale drawn on a paper to determine the level or intensity of pain in range of (0 to 10)
Goniometry | 3 months
  The science of measuring the joint ranges in each plane of the joint is called goniometry.
  Goniometer is a device that measures an angle or permits the rotation of an object to a definite position. Neck flexion, extension, side bending and rotation will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Manzoor, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Aziz Bhatti Shaheed hospital, Gujrat, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No